CLINICAL TRIAL: NCT00095706
Title: Phase I/II Combined Biological Therapy of Breast Cancer Using Monoclonal Antibodies Directed Against HER2/Neu Proto-Oncogene and Vascular Endothelial Growth Factor
Brief Title: Treatment of HER2-Positive Metastatic Breast Cancer With Herceptin and Bevacizumab (Antibodies Against HER2 and VEGF)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Translational Oncology Research International (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sara Hurvitz, University of California, Los Angeles
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TORI B-03; Western IRB #20041069; UCLA IRB #01-09-030; NCT00093535 (obsolete NCT alias)
Record Dates: First submitted 2004-11-05; First posted 2004-11-08 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer
Keywords: Metastatic breast cancer; HER2; Trastuzumab; Herceptin; VEGF; Bevacizumab; Avastin
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Pharmaceutical Preparations; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bevacizumab (drug), Herceptin (drug)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of combined treatment with trastuzumab (Herceptin) and bevacizumab (anti-VEGF antibody) in patients with HER2-positive metastatic breast cancer.

DETAILED DESCRIPTION:
Based on preclinical experiments conducted in our laboratories, we hypothesize that the aggressive behavior of HER2-overexpressing breast cancers is due in part to increased angiogenesis resulting from HER2-induced increases in vascular endothelial growth factor (VEGF) expression. In vivo experiments suggest that combined blockade of the HER2 receptor and VEGF results in superior anti-tumor efficacy compared with either treatment alone.

The current clinical trial, for which the phase I portion has been completed, will examine the efficacy and safety of trastuzumab (Herceptin) and bevacizumab (anti-VEGF antibody) in the treatment of HER2-overexpressing metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or relapsed locally advanced breast cancer
* HER2-positive by FISH
* No prior chemotherapy for metastatic disease
* ECOG performance status 0-2
* Normal left ventricular ejection fraction
* Bidimensionally measurable disease
* Oxygen saturation > 90% on room air

Exclusion Criteria:

* Other invasive malignancy within 5 years
* More than 3 different metastatic sites
* >50% liver involvement by metastasis
* Newly diagnosed untreated Stage IIIB breast cancer
* Prior chemotherapy for metastatic disease
* Clinically significant cardiovascular disease
* History or evidence of CNS disease
* Major surgery within 28 days prior to day 0
* Current or recent use of parenteral anticoagulants
* WBC < 3,000/uL
* Platelet count < 75,000/uL
* Hemoglobin < 9.0 g/dL
* Total Bilirubin > 2.0 mg/dL
* AST or ALT > 5 time upper limit of normal for subjects with documented liver metastases; > 2.5 times upper limit of normal for subjects without evidence of liver metastases
* Proteinuria (> 1g protein/24 hours at baseline)
* Prior therapy with Herceptin or rhuMAb VEGF (bevacizumab)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2003-06; Primary Completion 2007-04 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To establish the maximum tolerated dose (MTD) or recommended phase II dose of rhuMAb VEGF (bevacizumab) administered intravenously every 14 days to patients with HER2-amplified relapsed or metastatic breast cancer receiving concomitant Herceptin therapy

SECONDARY OUTCOMES:
To evaluate the clinical safety and toxicities of rhuMAb VEGF when administered in combination with Herceptin
To characterize the pharmacokinetics of rhuMAb VEGF and Herceptin given in combination
To evaluate the efficacy of rhuMAb VEGF plus Herceptin in terms of clinical activity when administered as an intravenous infusion, in patients with previously untreated metastatic or relapsed breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Pegram, MD, Principal Investigator — University of California, Los Angeles; Fairooz Kabbinavar, MD, Study Chair — Chief Medical Officer, TORI
Locations (18):
- United States (18):
  - Central Hematology Oncology Medical Group, Inc., Alhambra, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Virginia K. Crosson Cancer Center, Fullerton, California
  - Pacific Shores Medical Group, Long Beach, California
  - UCLA Medical Center, Los Angeles, California
  - North Valley Hematology/Oncology Medical Group, Northridge, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Wilshire Oncology Medical Group, Inc., Pomona, California
  - Cancer Care Associates Medical Group, Inc., Redondo Beach, California
  - Sansum Santa Barbara Medical Foundation Clinic, Santa Barbara, California
  - Santa Barbara Hematology Oncology Medical Group, Inc., Santa Barbara, California
  - San Diego Cancer Center, Vista, California
  - Cancer Institute of Florida, P.A., Orlando, Florida
  - Northeast Georgia Cancer Care, LLC, Athens, Georgia
  - Suburban Hematology-Oncology Associates, P.A., Lawrenceville, Georgia
  - Northwest Georgia Oncology Centers, P.C., Marietta, Georgia
  - Oncology Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada